CLINICAL TRIAL: NCT00307541
Title: Phase IIIa Randomized, Controlled Study to Assess the Immunogenicity of GlaxoSmithKline (GSK) Biologicals' 10-valent Pneumococcal Conjugate Vaccine, When Administered as a 3-dose Primary Immunization Course Before 6 Months of Age
Brief Title: Assess the Immunogenicity of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 105554; 2005-003299-40 (EudraCT Number)
Record Dates: First submitted 2006-03-07; First posted 2006-03-28 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae Vaccines
MeSH Terms: conditions — Streptococcal Infections | interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: Pneumococcal (vaccine)

SUMMARY:
Evaluate the immune response of GSK Biologicals' 10-valent pneumococcal conjugate vaccine one month after completion of a 3-dose primary vaccination course administered at 2, 3, 4 months of age

DETAILED DESCRIPTION:
Test groups: 2 groups (60 subjects/group). 10Pn-PD-DiT group receiving GSK Biologicals' 10-valent pneumococcal conjugate vaccine + DTPa-HBV-IPV/Hib; Control group receiving Prevenar + DTPa-HBV-IPV/Hib

ELIGIBILITY:
Inclusion criteria:

* Male or female between, and including, 8 and 16 weeks (56-118 days) of age at the time of the first vaccination, free of obvious health problems and with written informed consent obtained from the parent/guardian of the subject.

Exclusion criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a licensed vaccine not foreseen by the study protocol during the period starting from one month before the first dose of vaccine(s) and during the entire study period.

Ages: 8 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Start 2005-10-27 (Actual); Primary Completion 2006-04-07 (Actual); Study Completion 2006-04-07 (Actual)

PRIMARY OUTCOMES:
1 month post-dose 3: Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations >= 0.20 µg/mL

SECONDARY OUTCOMES:
1 month post dose 3: For all vaccine pneumococcal serotypes: Opsono titres
Antibody (Ab) concns >= 0.05 µg/mL
Ab concns to protein D and seropositivity (S+) status
S+/seroprotection status to antigens in DTPa-HBV-IPV/Hib vaccine
After each vaccination, occurrence of: solicited local, general symptoms within 4 days
Unsolicited adverse events within 31 days, SAEs (whole study period)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- Germany (26):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Marbach, Baden-Wurttemberg
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Tutzing, Bavaria
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Waren, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Gerolstein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Stollberg, Saxony
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=465

REFERENCES:
- [Background] Knuf M, Pankow-Culot H, Grunert D, Rapp M, Panzer F, Kollges R, Fanic A, Habib A, Borys D, Dieussaert I, Schuerman L. Induction of immunologic memory following primary vaccination with the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine in infants. Pediatr Infect Dis J. 2012 Jan;31(1):e31-6. doi: 10.1097/INF.0b013e3182323ac2. PMID 21909049
- See also: Booster Study — http://www.clinicaltrials.gov/ct/show/NCT00333450
- Available data/document: Study Protocol: 105554 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105554 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105554 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105554 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105554 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105554 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register